CLINICAL TRIAL: NCT04975295
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled, Multiple Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Subcutaneous LY3361237 in Participants With Psoriasis
Brief Title: A Study of LY3361237 in Participants With Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17291; I9S-MC-BTAC (Other: Eli Lilly and Company); 2019-003187-40 (EudraCT Number)
Record Dates: First submitted 2021-07-22; First posted 2021-07-23 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LY3361237 (Experimental): LY3361237 administered subcutaneously (SC).
  Interventions: Drug: LY3361237
- Placebo (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3361237 — Administered SC
  Arms: LY3361237
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to learn more about the safety and tolerability of LY3361237 and any side effects that might be associated with it when given to participants with psoriasis. LY3361237 will be administered by injections just under the skin. The study will last up to 41 weeks and may include up to 15 visits to the study center.

ELIGIBILITY:
Inclusion Criteria:

* Have chronic plaque psoriasis for at least 6 months
* Be willing and able to undergo skin biopsies
* Body mass index (BMI) within the range of 18 to 40 kilograms per meter squared (kg/m²)
* Female participants must agree to use birth control during the study

Exclusion Criteria:

* Have had certain types of infection within the last six months
* Have a clinically significant active infection, or recent acute active infection within the last 30 days
* Have other serious or unstable illnesses
* Have a history of organ or bone marrow transplant
* Have received any live vaccine within the last 4 weeks prior to screening
* Have received systemic nonbiologic psoriasis therapy within 4 weeks prior to study day 1
* Have received topical psoriasis treatment within 14 days prior to study day 1
* Have excessive skin exposure or use tanning booths for at least 4 weeks prior to study day 1

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment-Emergent Adverse Event(s) (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Day 253
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Minimum Serum Concentration (Cmin) of LY3361237 During the Dosing Interval | Day 1 predose through Day 253
  PK: Cmin of LY3361237 During the Dosing Interval

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- MC Comac Medical, Sofia, Bulgaria
- Budai Irgalmasrendi Korhaz, Budapest, Hungary
- Poland (4):
  - All Med - Lodz, Lodz
  - Ai Centrum Medyczne Sp. Z O.O. Sp.K., Poznan
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Pratia - Warsaw, Warsaw
- Summit Clinical Research, s.r.o. - Bratislava, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3361237 in Participants With Psoriasis — https://trials.lillytrialguide.com/en-US/trial/5M4E6fdkjelSDEBizWd8Bg